CLINICAL TRIAL: NCT06097442
Title: Effect of Apollo Wearable on Symptoms Related to Post-acute Sequelae SARS-CoV-2 Infection (PASC).
Brief Title: Effect of Apollo Wearable on Long COVID-19 Symptoms.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Board of Medicine (Other)
Collaborators: Apollo Neuroscience, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BOM0001
Record Dates: First submitted 2023-10-20; First posted 2023-10-24 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Post-acute Sequelae of SARS-COV-2 Infection
Keywords: long-COVID; Apollo
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Long-COVID Using Apollo: Participants with long-COVID symptoms who have consented to be part of this study will use an Apollo device according to a suggested schedule pre-set within their Apollo app, which participants can alter as they see fit.

SUMMARY:
The purpose of this study is to examine how Apollo wearable use impacts symptoms and quality of life following long COVID.

DETAILED DESCRIPTION:
Post-Acute Sequelae of SARS-CoV-2 infection (PASC), also known as long-COVID, is a syndrome that describes the persistence of symptoms or other sequelae weeks or months after initial SARS-CoV-2 infection. Limited evidence exists for effective treatments for this syndrome.

In this observational study, the investigators will examine the effects of Apollo wearable use on symptoms and quality of life related to long-COVID. The Apollo Neuroscience System (combined wearable and mobile application) offers a convenient, non-invasive, non-habit-forming wearable solution to improve performance and recovery under stress in children and adults. Our sample will be composed of new purchasers of Apollo or previous users of Apollo who haven't used Apollo in the preceding 14 days who are currently experiencing symptoms related to long-COVID according to PASC (self report).

Clinically validated survey tools will be administered upon enrollment in the study to assess baseline symptoms and quality of life. Once consented and enrolled in the study, participants will complete 7 monthly surveys for 6 months. Usage data from subjects' use of the wearable is also saved on the wearable directly and periodically uploaded to Apollo Neuroscience's secure and confidential database to be stored for analysis. Participants will first complete a screener survey to assess eligibility to participate. Demographic information and medication, substance, and treatment usage will also be collected.

Participants may choose to provide biometric data at their discretion for purposes of comparison at least 8 weeks before the study period, during the study period for 6 months, and at most 8 weeks after the study period. With regular Apollo use, the investigators expect to see an improvement in the physical, cognitive, and psychological symptoms associated with PASC. Initial analysis will compare subjects' baseline scores before Apollo use to scores during/after Apollo and the scores of subjects who used Apollo according to the study protocol and the scores of those who did not. Information gained from this study will help evaluate the use of Apollo as a potential non-invasive and accessible solution to aid in reducing long-COVID symptoms.

ELIGIBILITY:
Inclusion Criteria:

* New purchasers of Apollo who haven't started using their Apollo device or previous users of Apollo who haven't used Apollo in the preceding 14 days.
* Age 18 years or over
* Currently experiencing symptoms related to long-COVID according to PASC (self report).
* Must be experiencing PASC symptoms in at least one of the following domains:

Respiratory-related symptoms Fatigue-related symptoms Neurologic-related symptoms Psychiatric-related symptoms Sleep-related symptoms Change in quality of life/functional status

Exclusion Criteria:

* Inability to use or access a compatible Android or iOS smartphone
* Are unable to complete consent and questionnaires written in English
* Current resident of a European Union (EU) country

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Existing or new customers of Apollo Neuro wellness device
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Post-Covid-19 Functional Status Scale (PCFS) | Monthly for 6 months
  Post-Covid-19 Functional Status Scale (PCFS) will be used to assess participants' functional recovery following a COVID-19 diagnosis.

SECONDARY OUTCOMES:
Modified Medical Research Council (mMRC) Dyspnea Scale | Monthly for 6 months
  The Modified Medical Research Council (mMRC) Dyspnea Scale will be used to assess dyspnea (labored breathing).
EuroQol-5D-5L (EQ-5D) | Monthly for 6 months
  The EuroQol-5D-5L (EQ-5D) will measure health in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Neurobehavioral Symptom Inventory (NSI) | Monthly for 6 months
  The Neurobehavioral Symptom Inventory (NSI) will be used to assess neurobehavioral symptoms.
Fatigue Severity Scale (FSS) | Monthly for 6 months
  The Fatigue Severity Scale (FSS) will be used to measure the severity of fatigue symptoms.
Pittsburgh Sleep Quality Index (PSQI) | Monthly for 6 months
  The Pittsburgh Sleep Quality Index (PSQI) will be used to quantify sleep quality and disturbances over a month interval at a time.

CONTACTS AND LOCATIONS:
Locations (1):
- The Board of Medicine, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No